CLINICAL TRIAL: NCT02083393
Title: Changes of Dendritic Cells in Acute Lung Injury
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Zhongda Hospital, Southeast University, China
Other Study IDs: SoutheastUChina2011ZDllKY04
Record Dates: First submitted 2011-09-28; First posted 2014-03-11 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Acute Lung Injury
Keywords: dendritic cell
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with acute lung injury: Patients with sepsis induced acute lung injury
- Postsurgery patients: Postsurgery patients without acute lung injury and sepsis

SUMMARY:
To observe changes of circulating and tissue dendritic cells in acute lung injury,including invasive aspergillosis pneumonia

DETAILED DESCRIPTION:
Change of circulating and tissular dendritic cells of patients with acute lung injury was still unclear, we used a flow cytometry-based assay to quantify circulating and tissular DCs and their HLA-DR surface expression at the time of diagnosis and during the first week of evolution in patients with acute lung injury, and healthy people as controls.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis induced acute lung injury

Exclusion Criteria:

* Younger than 18-year-old
* Pregnancy
* Cancer or organ transplant
* Asthma
* COPD
* Heart Failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sepsis induced-ALI patients with mechanical ventilation including invasive aspergillosis
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2011-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28day

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Qiu, Ph.D., Principal Investigator — Southeast University
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China